CLINICAL TRIAL: NCT05622331
Title: Burden of Respiratory Syncytial Virus (RSV) in Children in Sweden (BRICS): A Retrospective Study in Sweden
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: Quantify Research (Unknown)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: RSV00046; U1111-1280-4878 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-10-28; First posted 2022-11-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- RSV cohort: Children (<5 years of age at diagnosis) with a diagnosis of RSV (ICD-10 code) in hospital care between July 1st 2006 and June 30th 2021
- Regional primary care RSV cohort: Children (<5 year of age) with a diagnosis of RSV (ICD-10 code) in primary care identified in regional databases (Region Skåne, Region Halland and VGR) between July 1st 2006 and June 30th 2021
- Regional laboratory RSV cohort: Children (<5 years of age) with a positive laboratory RSV test result (multiplex/rapid PCR, antigen, immunofluorescence or immunochromatography rapid test) in primary or hospital care, identified in regional laboratory databases (Region Skåne and Region Halland) between July 1st 2006 and June 30th 2021
- Acute Respiratory Infections (ARI) cohort: Children (<5 of age) with a diagnosis of ARI (ICD-10 code,) in hospital care between July 1st 2006 and June 30th 2021
- Regional ARI cohort: Children (<5 years of age) with a diagnosis of RSV (ICD-10 code, see Table 1) in primary care, identified in regional databases (Region Skåne, Region Halland and VGR)
- Rhinovirus cohort: Children (<5 of age) with a diagnosis of rhinovirus (ICD-10 code,) in hospital care between July 1st 2006 and June 30th 2021
- Human Metapneumovirus (HMPV) cohort: Children (<5 of age) with a diagnosis of HMPV (ICD-10 code,) in hospital care between July 1st 2006 and June 30th 2021
- Parainfluenza cohort: Children (<5 of age) with a diagnosis of parainfluenza (ICD-10 code,) in hospital care between July 1st 2006 and June 30th 2021
- Parent cohort: Parents to all children will be linked to the study population, which is possible through linkage between children and parents by their personal identifiers
- Non-RSV control cohort: A non-RSV control population consisting of children (<5 years of age) will be extracted to estimate the burden compared to the general population

SUMMARY:
Primary Objective:

-Estimate the hospital-associated healthcare resource use (HCRU), and associated costs, of RSV infection in children in comparison to the non-RSV control cohort (general population) and patients with rhinovirus infection.

Secondary Objectives:

* Describe demographic and clinical patient characteristics of RSV infected children.
* Estimate and compare the incidence of RSV infection and acute respiratory infections (ARIs) in children.
* Estimate the mortality associated with RSV infection in children.
* Estimate the social economic burden of RSV infection in children in relation to parents staying home from work to care for their sick child (VAB leave) in comparison to non-RSV control cohort (i.e. parents to children in the general population).

  * Estimate the net days with VAB leave and the compensation disbursed (temporary parental benefit) associated with RSV infection in children.
  * Estimate the indirect costs that can be attributed to VAB leave.
* Examine the medium- and long-term complications associated with an RSV diagnosis in children in comparison to the non-RSV control chart (general population) and patients with rhinovirus infection.
* Examine and describe risk factors associated with an RSV infection in children
* Estimate the healthcare resource use (HCRU), and associated costs, of RSV infection in children, for a subset of patients where primary care data is available, in comparison to the non-RSV control cohort (general population).

DETAILED DESCRIPTION:
The overall study period will be between July 1st 2001 and to latest available date (likely June 30th 2022).

Patients will be identified for inclusion in the study population between July 1st 2006 and June 30th 2021.

Patients will be followed from time of inclusion until end of the study period or until death.

All patients will have an index date corresponding to the date of diagnosis of incident infection in primary and/or hospital care during the identification period. An incident infection is defined as the occurrence of infections more than 30 (>30) days apart. This implies that a patient can have more than one index date during the study period. Patients that are included in both the RSV cohort and the regional primary care RSV cohort may have two different index dates for the same incident infection, depending on the objective. This is if a patient is first treated in primary care and then hospitalized. The index date is defined differently for the two cohorts, as the first diagnosis in hospital care for the RSV cohort and first diagnosis in primary care OR hospital care for the regional primary care cohort. The non-RSV controls will have the same index date as their matched RSV patient.

The look-back period will be used to inform baseline characteristics as well as patients' medical and diagnosis history. All patients will have possible look-back from birth for information on the patient's hospital care history and from 2005 for information on the patient's prescribed drugs history. The individual look-back and follow-up will depend on the time of inclusion in the study population as well as age at inclusion.

ELIGIBILITY:
Inclusion Criteria:

•Children (≤5 years of age) with an RSV infection or any acute respiratory infection (ARI) between July 1st 2001 and latest available date, identified in either hospital care, regional primary care or laboratory database.

Exclusion Criteria:

•There are no exclusion criteria for this study.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The source population for this study will consist of all children (≤5 years of age) in Sweden with an RSV infection or any acute respiratory infection (ARI) between January 1rst 2001 and latest available date, identified from three sources:
  * Primary or secondary diagnosis in hospital care (National Patient Registry)
  * Primary or secondary diagnosis in primary care (regional databases)
  * Positive RSV laboratory test result (Regional laboratory data) The expected study sample is 38,000 unique pediatric patients with an RSV diagnosis, identified in the National Patient Register between 2001 and 2020. The expected RSV sample size, the non-RSV control population will consist of 80,000-160,000 individuals, matched 1:10. The expected number of ARI infections during the time period is estimated to around 1 million. This totals a study sample of between 1-1.1 million.
Sampling Method: Non-Probability Sample
Enrollment: 1100000 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Short-term healthcare: Number of specialist outpatient visits | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  Number of RSV specialist outpatient hospital visits during follow-up
Short-term healthcare: Number of hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  Number of hospitalizations/stays related to RSV during follow-up
Short-term healthcare: Length of hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  The length of hospitalizations/stays related to RSV during follow-up
Short-term healthcare: Number of Intensive Care Unit (ICU) hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  Number of ICU hospitalizations/stays related to RSV during follow-up
Short-term healthcare: Length of ICU hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  The length of ICU hospitalizations/stays related to RSV during follow-up
Short-term healthcare: Number of RSV-related medical/surgical procedures | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  Number of RSV-related medical/surgical procedures during follow-up
Short-term healthcare: Number of dispensed prescriptions of RSV-related medications | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  Number of dispensed prescriptions of RSV-related medications during follow-up
Short-term healthcare: The costs of direct medical (in- and outpatient care) | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  Direct medical (in- and outpatient care) costs related to RSV infection
Short-term healthcare: The costs of RSV-related medications | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  The costs of dispensed prescriptions of RSV-related medications based on pharmacy retail price
Medium-term healthcare: Number of specialist outpatient visits | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Number of RSV specialist outpatient hospital visits during follow-up
Medium-term healthcare: Number of hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Number of hospitalizations/stays related to RSV during follow up
Medium-term healthcare: Length of hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  The length of hospitalizations/stays related to RSV during follow up
Medium-term healthcare: Number of Intensive Care Unit (ICU) hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Number of ICU hospitalizations/stays related to RSV during follow-up
Medium-term healthcare: Length of ICU hospitalizations | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  The length of ICU hospitalizations/stays related to RSV during follow-up
Medium-term healthcare: Number of RSV-related medical/surgical procedures | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Number of RSV-related medical/surgical procedures during follow-up
Medium-term healthcare: Number of dispensed prescriptions of RSV-related medications | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Number of dispensed prescriptions of RSV-related medications during follow-up
Medium-term healthcare: The costs of direct medical (in- and outpatient care) | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Direct medical (in- and outpatient care) costs related to RSV infection
Medium-term healthcare: The costs of RSV-related medications | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  The costs of dispensed prescriptions of RSV-related medications based on pharmacy retail price

SECONDARY OUTCOMES:
Patient characteristics | Analysis period: July 1st 2006 - June 30th 2021 Reporting period: at index date or during look-back period
  Age at diagnosis, sex distribution, region of residence, birth weight, birth height, gestational age, mothers age at birth, high-risk conditions, parent's education, parent's income, household status
Incidence of RSV/ARIs | Analysis period: July 1st 2006 - June 30th 2021 Reporting period: by respiratory years
  Incidence of RSV/ARI per 100,000 population
Number of laboratory-confirmed RSV cases with RSV diagnosis | Analysis period: July 1st 2006 - June 30th 2021 Reporting period: at index date or during look-back period
  Number of laboratory confirmed RSV cases with RSV diagnosis code (ICD-10)
Number of laboratory-confirmed RSV cases with no RSV diagnosis | Analysis period: July 1st 2006 - June 30th 2021Reporting period: at index date or during look-back period
  Number of laboratory confirmed RSV cases with no RSV diagnosis code (ICD-10)
Number of diagnosed RSV cases with no RSV laboratory tests conducted | Analysis period: July 1st 2006 - June 30th 2021 Reporting period: at index date or during look-back period
  Number of diagnosed RSV cases (ICD-10) with no laboratory test conducted
Mortality | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 30 days from index date
  All-cause 30-day death from index date
Socioeconomic burden: Net days of VAB leave | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Net days of temporary parental leave (VAB) during follow-up period due to child with RSV diagnosis
Socioeconomic burden: Net VAB leave benefit | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Net temporary parental leave (VAB) benefit during follow-up period due to child with RSV diagnosis
Socioeconomic burden: Indirect costs of VAB leave due to RSV | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: 12 months from (first) index date
  Productivity loss due to RSV-related temporary parental leave during follow-up period, calculated by human capital method and average wage
Proportion of patients that develop respiratory complications (ICD-10 codes) | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: per year during 5 years from index date
  Proportion of patients that develop respiratory complications (ICD-10 codes)
Incidence of RSV per 1000 person-years | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: per year during 5 years from index date
  Incidence of RSV per 1000 person-years in RSV, non-RSV control cohorts and rhinovirus cohorts
Incidence rate ratios (IRR) | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: per year during 5 years from index date
  Incidence rate ratios (IRR) in RSV, non-RSV control and rhinovirus cohorts
Hazard ratios (HR) | Analysis period: July 1st 2006 - July 31st 2021 Reporting period: per year during 5 years from index date
  Hazard ratios (HR) in RSV, non-RSV control and rhinovirus cohorts
Estimation of hazard ratio of each risk factor on being diagnosed with RSV | Analysis period: July 1st 2006 - July 31st 2021Reporting period: look back period
  A Cox proportional hazards regression model will be used to estimate the hazard ratio of each risk factor on being diagnosed with RSV. Predictors for RSV diagnosis presented as hazard ratios, including premature birth, high-risk conditions, APGAR, seasonality, mother's age at birth, number of children in household, birth order, parent's education, parent's income, household status, maternal smoking, mother's BMI
Primary Care: Number of primary care contacts | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Number of primary care contacts during follow-up period
Primary Care: Number of specialized outpatient care visits | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Number of specialized outpatient care visits during follow-up period
Primary Care: Number of hospitalizations | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Number of hospitalizations/stays related to RSV during follow-up
Primary Care: Length of hospitalizations | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Length of hospitalizations/stays related to RSV during follow-up
Primary Care: Number of ICU hospitalizations | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Number of ICU hospitalizations/stays related to RSV during follow-up
Primary Care: Length of ICU hospitalizations | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Length of ICU hospitalizations/stays related to RSV during follow-up
Primary Care: Number of RSV-related medical/surgical procedures | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Number of RSV-related medical/surgical procedures during follow-up
Primary Care: Number of dispensed prescriptions of RSV-related medications | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Number of dispensed prescriptions of RSV-related medications during follow-up
Primary Care: The costs of direct medical (in- and outpatient care) | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  Direct medical (in- and outpatient care) costs related to RSV infection
Primary Care: The costs of RSV-related medications | Analysis period: Date of first available data - July 31st 2021 Reporting period: 30 days from index date
  The costs of dispensed prescriptions of RSV-related medications based on pharmacy retail price

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org